CLINICAL TRIAL: NCT03938636
Title: Evaluation of the Precision and Sensitivity of Tilmanocept Uptake Value (TUV) on Tc 99m Tilmanocept Planar Imaging
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Navidea Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NAV3-31
Record Dates: First submitted 2019-04-24; First posted 2019-05-06 (Actual); Results first posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Rheumatoid Arthritis
Keywords: RA; healthy control; tilmanocept; diagnostic; imaging
MeSH Terms: conditions — Arthritis, Rheumatoid; Disease | interventions — technetium-diethylenetriaminepentaacetic acid-mannosyl-dextran

STUDY DESIGN:
Intervention Model Description: This is a prospective, open-label, multicenter, single and repeated-dose study designed to evaluate the reliability and sensitivity of TUV assessments in healthy controls and subjects with active RA.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Subjects free of inflammatory disease (Experimental): Arm 1 includes inflammatory-disease-free HCs. Arm 1 was designed to evaluate image/re-image consistency (repeatability and stability) of joint-specific and global TUVs across a variety of image acquisition intervals and to collect normative HC data.
  Interventions: Drug: Tc 99m tilmanocept
- RA subjects on stable therapy (Experimental): Arm 2 includes clinically-diagnosed RA subjects on stable treatment. Arm 2 was designed to evaluate image/re-image and test re-test (i.e., repeated dose) consistency of joint-specific and global TUVs across a variety of image acquisition intervals.
  Interventions: Drug: Tc 99m tilmanocept
- RA subjects who are candidates for initiation of a new anti-TNFα therapy (Experimental): Arm 3 includes clinically-diagnosed RA subjects on stable treatment who are candidates for initiation of, or change to, new anti-TNFα therapy. Arm 3 was designed to assess the efficacy of global TUVs, obtained before and after initiation of a new anti-TNFα therapy, to predict future clinical responsiveness to the new therapy.
  Interventions: Drug: Tc 99m tilmanocept

INTERVENTIONS:
Drug: Tc 99m tilmanocept — Tilmanocept is a radiotracer that accumulates in macrophages by binding to a mannose binding receptor that resides on the surface.
  Other Names: Lymphoseek

SUMMARY:
This clinical trial will look at scans of the hands and wrists taken from healthy control subjects (HCs) and from subjects with rheumatoid arthritis (RA). Before each scan, subjects will be given an injection of Tc 99m tilmanocept to help the scan identify inflammation in the hand and wrist joints, which can be a part of the RA disease. Data from the scans will be used to calculate a number referred to as tilmanocept uptake value (or TUV) that is a measure of how much Tc 99m tilmanocept has located in the joints. The questions this trial aims to answer are:

* How consistent are the scan results (TUVs) when the scans are repeated over time?
* What are normal TUVs in healthy people? This will help define abnormally high values in people with RA.
* Are TUVs calculated early after a person starts a new drug to treat RA able to predict whether that person will have a good response to the drug later on (after it has had time to take full effect several weeks later)?

DETAILED DESCRIPTION:
This trial is a prospective, open-label, multicenter, single and repeated-dose study designed to evaluate the reliability and sensitivity of TUV assessments in healthy control subjects and subjects with active RA.

This study is stratified into 3 arms. The first 2 arms, consisting of [1] disease-free HCs and [2] clinically diagnosed RA subjects on stable treatment, respectively, are designed to evaluate the image re-image and/or test re-test (i.e., repeated dose) consistency of joint-specific and global TUVs across a variety of image acquisition intervals.

The third arm consists of clinically-diagnosed subjects with active RA who are candidates for initiation of, or change to, a new anti-TNFα bDMARD therapy. This arm is designed to assess the efficacy of TUVglobal as an early predictor of response to the new anti-TNFα bDMARD therapy.

ELIGIBILITY:
Inclusion Criteria:

ALL SUBJECTS:

1. The subject has provided written informed consent with HIPAA (Health Information Portability and Accountability Act) authorization before the initiation of any study-related procedures.
2. ARMS 1 and 2 (only): The subject has agreed to not engage in any diet, lifestyle, or medication changes until study completion.

   HEALTHY CONTROL SUBJECTS
3. The subject is between 18 and 80 years of age at the time of consent.
4. The subject is deemed to be clinically free of any inflammatory disease(s) and has not experienced joint pain for at least 28 days prior to the consent date.
5. The subject is not currently on anti-inflammatory drugs (including NSAIDs) and has not taken anti-inflammatories for at least 28 days prior to the consent date.
6. For all ongoing concomitant medications, the subject has maintained a stable dose for at least 28 days prior to the consent date.

CLINICALLY DIAGNOSED ACTIVE RA SUBJECTS:

3. The subject is at least 18 years of age and was ≥ 18 years of age at the time of RA diagnosis.

4. The subject has moderate to severe RA as determined by the 2010 American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) Classification Criteria (score of ≥ 6/10).

5. The subject has a 28-joint disease activity score (DAS28) of ≥ 3.2 (includes the Erythrocyte Sedimentation Rate [ESR] test and Visual Analog Scale [VAS]).

6. Subjects receiving traditional DMARDs must have been on therapy for ≥ 90 days and at a stable dose for ≥ 30 days prior to the first imaging visit (Day 0).

7. If the subject is receiving bDMARD or janus kinase (JAK) inhibitor therapy, they have been at a stable dose > 180 days prior to the first imaging visit (Day 0).

8. If the subject is receiving NSAIDs or oral corticosteroids, the dose has been stable for > 28 days prior to first imaging visit (Day 1). The corticosteroid dose must be ≤ 10 mg/day of prednisone or an equivalent steroid dose.

9. ARM 3 (only): The subject is receiving anti-rheumatic treatment and is a candidate for initiation of, or change to, a new anti-TNFα bDMARD treatment.

Exclusion Criteria:

1. The subject is pregnant or lactating.
2. The subject size or weight is not compatible with imaging per the investigator.
3. The subject has had or is currently receiving radiation therapy or chemotherapy.
4. The subject has renal insufficiency as demonstrated by a glomerular filtration rate of < 60 mL/min.
5. The subject has hepatic insufficiency as demonstrated by ALT (alanine aminotransferase [SGPT]) or AST (aspartate aminotransferase [SGOT]) greater than 3 times the upper limit of normal.
6. The subject has any severe, acute, or chronic medical conditions and/or psychiatric conditions and/or laboratory abnormalities that would impart, in the judgment of the investigator, excess risk associated with study participation or study drug administration that would deem the subject inappropriate for study participation.
7. The subject has a known allergy to or has had an adverse reaction to dextran exposure.
8. The subject has received an investigational product within 30 days prior to the Tc 99m tilmanocept administration.
9. The subject has received intra-articular corticosteroid injections ≤ 8 weeks prior to the first imaging visit (Day 0).
10. The subject has received any radiopharmaceutical within 7 days or 10 half-lives prior to the administration of Tc 99m tilmanocept.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2021-02-08 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Blue, MD, Study Director — Navidea Biopharmaceuticals
Locations (10):
- United States (10):
  - Imaging Endpoints, Scottsdale, Arizona
  - Axis Clinical Trials, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - Innovation Medical Research Center, Palmetto Bay, Florida
  - Physician Research Collaboration, Lincoln, Nebraska
  - University Hospitals, Cleveland, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Central States Research, Tulsa, Oklahoma
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Subjects Free of Inflammatory Disease: Arm 1 comprises disease-free HCs. Arm 1 was designed to evaluate image/re-image consistency (repeatability and stability) of joint-specific and global TUVs across a variety of image acquisition intervals and to collect normative HC data.
  TC99m-tilmanocept: Tilmanocept is a radiotracer that accumulates in macrophages by binding to a mannose binding receptor that resides on the surface.
- RA Subjects on Stable Therapy: Arm 2 comprises clinically diagnosed RA subjects on stable treatment. Arm 2 was designed to evaluate image/re-image and test re-test (i.e., repeat dose) consistency of joint-specific and global TUVs across a variety of image acquisition intervals.
  TC99m-tilmanocept: Tilmanocept is a radiotracer that accumulates in macrophages by binding to a mannose binding receptor that resides on the surface.
- Candidates for Initiation of a New Anti-TNFα Therapy: Arm 3 comprises clinically diagnosed RA subjects on stable treatment who are candidates for initiation of, or change to, new anti-TNFα therapy. Arm 3 was designed to assess the efficacy of global TUVs, obtained before and after initiation of a new anti-TNFα therapy, to predict future clinical responsiveness to the new therapy.
  TC99m-tilmanocept: Tilmanocept is a radiotracer that accumulates in macrophages by binding to a mannose binding receptor that resides on the surface.
Period: Overall Study
Arm/Group | Subjects Free of Inflammatory Disease | RA Subjects on Stable Therapy | Candidates for Initiation of a New Anti-TNFα Therapy
Started | 44 | 41 | 31
Completed | 44 (15 Arm 1 subjects were deemed non-evaluable due to image acquisition and image quality deviations.) | 38 | 28
Not Completed | 0 | 3 | 3
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Subject withdrew due to death in family | 0 | 1 | 0
Not completed — Missed visit | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Subjects Free of Inflammatory Disease: Arm 1 comprised disease-free HCs. Arm 1 evaluated image/re-image consistency (repeatability and stability) of joint-specific and global TUVs across a variety of image acquisition intervals and collect normative HC data.
  Tc99m-tilmanocept: Tilmanocept is a radiotracer that accumulates in macrophages by binding to a mannose binding receptor that resides on the surface.
- RA Subjects on Stable Therapy: Arm 2 comprised clinically diagnosed RA subjects on stable treatment. Arm 2 evaluated image/re-image and test re-test (i.e., repeat dose) consistency of joint-specific and global TUVs across a variety of image acquisition intervals.
  Tc99m-tilmanocept: Tilmanocept is a radiotracer that accumulates in macrophages by binding to a mannose binding receptor that resides on the surface.
- RA Subjects Who Are Candidates for Initiation of a New Anti-TNFα Therapy: Arm 3 comprised clinically diagnosed RA subjects on stable treatment who were candidates for new anti-TNFα therapy. Arm 3 assessed the efficacy of global TUVs, obtained before and after initiation of a new anti-TNFα therapy, to predict future clinical responsiveness to the new therapy.
  Tc99m-tilmanocept: Tilmanocept is a radiotracer that accumulates in macrophages by binding to a mannose binding receptor that resides on the surface.
- Total: Total of all reporting groups
Arm/Group | Subjects Free of Inflammatory Disease | RA Subjects on Stable Therapy | RA Subjects Who Are Candidates for Initiation of a New Anti-TNFα Therapy | Total
Number analyzed (Participants) | 44 | 41 | 31 | 116
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 44 | 31 | 22 | 97
  >=65 years | 0 | 10 | 9 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.8 (10.98) | 56.8 (11.19) | 57.0 (13.68) | 49.3 (15.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 34 | 25 | 85
  Male | 18 | 7 | 6 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 3 | 15 | 31
  Not Hispanic or Latino | 31 | 38 | 16 | 85
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 2 | 2 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 17 | 11 | 2 | 30
  White | 24 | 23 | 28 | 75
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 4 | 0 | 5
Region of Enrollment [Number; unit: participants]
  United States | 44 | 41 | 31 | 116

OUTCOME MEASURES:

1. Primary Outcome: Arms 1 & 2: Assess Camera-specific Precision of TUV
Description: The camera-specific precision of TUVjoint in subjects with active RA and Healthy Controls (HCs), which is described as the Root Mean Square Difference (RMSD) between the 15-minute planar images (referred to as A and B images at 60 and 180 minutes). The RMSD is calculated as the square root of the mean squared deviation from zero.
Time Frame: Day 0 tilmanocept injection followed by imaging at 60 minutes (60A) and 75 minutes (60B) and at 180 minutes (180A) and 195 minutes (180B).
Population: Planned interim analysis of first 15 subjects in Arms 1 and 2
Measure: Number (95% Confidence Interval); unit: Pixel intensity
Arm/Group | Subjects Free of Inflammatory Disease | RA Subjects on Stable Therapy
Number analyzed (Participants) | 15 | 15
Pixel intensity
  Left metacarpophalangeal 1, RMSD of TUV at 60 min A vs 60 min B | 0.159 [0.11 to 0.23] | 0.067 [0.05 to 0.10]
  Left metacarpophalangeal 2, RMSD of TUV at 60 min A vs 60 min B | 0.091 [0.07 to 0.14] | 0.124 [0.09 to 0.19]
  Left metacarpophalangeal 3, RMSD of TUV at 60 min A vs 60 min B | 0.087 [0.06 to 0.13] | 0.125 [0.09 to 0.19]
  Left metacarpophalangeal 4, RMSD of TUV at 60 min A vs 60 min B | 0.094 [0.07 to 0.14] | 0.130 [0.09 to 0.20]
  Left metacarpophalangeal 5, RMSD of TUV at 60 min A vs 60 min B | 0.077 [0.06 to 0.12] | 0.070 [0.05 to 0.09]
  Left proximal interphalangeal 1, RMSD of TUV at 60 min A vs 60 min B | 0.078 [0.05 to 0.11] | 0.080 [0.05 to 0.10]
  Left proximal interphalangeal 2, RMSD of TUV at 60 min A vs 60 min B | 0.058 [0.04 to 0.09] | 0.066 [0.05 to 0.10]
  Left proximal interphalangeal 3, RMSD of TUV at 60 min A vs 60 min B | 0.064 [0.05 to 0.10] | 0.099 [0.07 to 0.14]
  Left proximal interphalangeal 4, RMSD of TUV at 60 min A vs 60 min B | 0.080 [0.06 to 0.12] | 0.077 [0.05 to 0.11]
  Left proximal interphalangeal 5, RMSD of TUV at 60 min A vs 60 min B | 0.050 [0.03 to 0.07] | 0.043 [0.03 to 0.07]
  Left wrist, RMSD of TUV at 60 min A vs 60 min B | 0.089 [0.06 to 0.13] | 0.086 [0.06 to 0.13]
  Right metacarpophalangeal 1, RMSD of TUV at 60 min A vs 60 min B | 0.124 [0.08 to 0.17] | 0.083 [0.05 to 0.11]
  Right metacarpophalangeal 2, RMSD of TUV at 60 min A vs 60 min B | 0.096 [0.07 to 0.14] | 0.165 [0.12 to 0.25]
  Right metacarpophalangeal 3, RMSD of TUV at 60 min A vs 60 min B | 0.097 [0.07 to 0.15] | 0.152 [0.11 to 0.23]
  Right metacarpophalangeal 4, RMSD of TUV at 60 min A vs 60 min B | 0.058 [0.04 to 0.09] | 0.069 [0.05 to 0.10]
  Right metacarpophalangeal 5, RMSD of TUV at 60 min A vs 60 min B | 0.067 [0.05 to 0.10] | 0.062 [0.05 to 0.10]
  Right proximal interphalangeal 1, RMSD of TUV at 60 min A vs 60 min B | 0.090 [0.06 to 0.14] | 0.095 [0.07 to 0.14]
  Right proximal interphalangeal 2, RMSD of TUV at 60 min A vs 60 min B | 0.080 [0.06 to 0.12] | 0.070 [0.05 to 0.11]
  Right proximal interphalangeal 3, RMSD of TUV at 60 min A vs 60 min B | 0.062 [0.05 to 0.10] | 0.059 [0.04 to 0.09]
  Right proximal interphalangeal 4, RMSD of TUV at 60 min A vs 60 min B | 0.084 [0.06 to 0.12] | 0.095 [0.07 to 0.14]
  Right proximal interphalangeal 5, RMSD of TUV at 60 min A vs 60 min B | 0.048 [0.04 to 0.07] | 0.111 [0.08 to 0.17]
  Right wrist 5, RMSD of TUV at 60 min A vs 60 min B | 0.070 [0.05 to 0.10] | 0.097 [0.07 to 0.15]
  Left metacarpophalangeal 1, RMSD of TUV at 180 min A vs 180 min B | 0.119 [0.09 to 0.18] | 0.113 [0.08 to 0.17]
  Left metacarpophalangeal 2, RMSD of TUV at 180 min A vs 180 min B | 0.086 [0.06 to 0.13] | 0.167 [0.11 to 0.23]
  Left metacarpophalangeal 3, RMSD of TUV at 180 min A vs 180 min B | 0.090 [0.06 to 0.14] | 0.097 [0.07 to 0.14]
  Left metacarpophalangeal 4, RMSD of TUV at 180 min A vs 180 min B | 0.110 [0.07 to 0.14] | 0.106 [0.08 to 0.16]
  Left metacarpophalangeal 5, RMSD of TUV at 180 min A vs 180 min B | 0.097 [0.06 to 0.13] | 0.114 [0.08 to 0.18]
  Left proximal interphalangeal 1, RMSD of TUV at 180 min A vs 180 min B | 0.071 [0.04 to 0.09] | 0.106 [0.08 to 0.16]
  Left proximal interphalangeal 2, RMSD of TUV at 180 min A vs 180 min B | 0.050 [0.03 to 0.07] | 0.075 [0.05 to 0.11]
  Left proximal interphalangeal 3, RMSD of TUV at 180 min A vs 180 min B | 0.057 [0.04 to 0.08] | 0.131 [0.09 to 0.20]
  Left proximal interphalangeal 4, RMSD of TUV at 180 min A vs 180 min B | 0.068 [0.05 to 0.10] | 0.083 [0.06 to 0.13]
  Left proximal interphalangeal 5, RMSD of TUV at 180 min A vs 180 min B | 0.077 [0.05 to 0.10] | 0.073 [0.05 to 0.11]
  Left wrist, RMSD of TUV at 180 min A vs 180 min B | 0.085 [0.05 to 0.11] | 0.137 [0.09 to 0.18]
  Right metacarpophalangeal 1, RMSD of TUV at 180 min A vs 180 min B | 0.079 [0.06 to 0.12] | 0.109 [0.08 to 0.16]
  Right metacarpophalangeal 2, RMSD of TUV at 180 min A vs 180 min B | 0.097 [0.07 to 0.15] | 0.184 [0.13 to 0.27]
  Right metacarpophalangeal 3, RMSD of TUV at 180 min A vs 180 min B | 0.083 [0.06 to 0.13] | 0.138 [0.10 to 0.20]
  Right metacarpophalangeal 4, RMSD of TUV at 180 min A vs 180 min B | 0.103 [0.07 to 0.14] | 0.105 [0.08 to 0.16]
  Right metacarpophalangeal 5, RMSD of TUV at 180 min A vs 180 min B | 0.076 [0.05 to 0.10] | 0.078 [0.06 to 0.12]
  Right proximal interphalangeal 1, RMSD of TUV at 180 min A vs 180 min B | 0.065 [0.05 to 0.09] | 0.107 [0.07 to 0.14]
  Right proximal interphalangeal 2, RMSD of TUV at 180 min A vs 180 min B | 0.086 [0.06 to 0.13] | 0.088 [0.06 to 0.13]
  Right proximal interphalangeal 3, RMSD of TUV at 180 min A vs 180 min B | 0.056 [0.04 to 0.08] | 0.125 [0.09 to 0.19]
  Right proximal interphalangeal 4, RMSD of TUV at 180 min A vs 180 min B | 0.048 [0.03 to 0.07] | 0.099 [0.07 to 0.15]
  Right wrist, RMSD of TUV at 180 min A vs 180 min B | 0.087 [0.06 to 0.11] | 0.163 [0.11 to 0.22]

2. Primary Outcome: Arms 1 and 2: Stability of the Mean/Variance Relationship
Description: The stability of the mean/variance relationship, which is assessed by comparing the Coefficient of Variation (CV) of TUVjoint and TUVglobal in subjects with active RA and in healthy control subjects at 60 and 180 minutes.
Time Frame: Day 0 tilmanocept injection followed by imaging at 60 minutes and 180 minutes.
Population: Planned interim analysis of first 15 subjects in Arms 1 and 2
Measure: Number; unit: Coefficient of variation
Arm/Group | Subjects Free of Inflammatory Disease | RA Subjects on Stable Therapy
Number analyzed (Participants) | 15 | 15
Coefficient of variation
  Global TUV at 60 min: number analyzed (Participants) | 15 | 9
  Global TUV at 60 min | 263.31 | 208.79
  Left metacarpophalangeal 1 TUV at 60 min | 16.92295 | 13.189704
  Left metacarpophalangeal 2 TUV at 60 min | 19.613096 | 20.477108
  Left metacarpophalangeal 3 TUV at 60 min | 18.651035 | 16.378147
  Left metacarpophalangeal 4 TUV at 60 min | 18.511573 | 13.970308
  Left metacarpophalangeal 5 TUV at 60 min | 21.20135 | 12.21378
  Left proximal interphalangeal 1 TUV at 60 min | 12.819593 | 11.370952
  Left proximal interphalangeal 2 TUV at 60 min | 17.553684 | 9.7087077
  Left proximal interphalangeal 3 TUV at 60 min | 17.847881 | 12.604637
  Left proximal interphalangeal 4 TUV at 60 min | 17.407371 | 15.660407
  Left proximal interphalangeal 5 TUV at 60 min | 14.424961 | 10.066291
  Left wrist TUV at 60 min | 14.401304 | 8.7901247
  Right metacarpophalangeal 1 TUV at 60 min | 13.628956 | 11.48462
  Right metacarpophalangeal 2 TUV at 60 min | 19.774959 | 18.014491
  Right metacarpophalangeal 3 TUV at 60 min | 20.228576 | 23.49369
  Right metacarpophalangeal 4 TUV at 60 min | 18.728588 | 18.207621
  Right metacarpophalangeal 5 TUV at 60 min | 19.283062 | 12.958136
  Right proximal interphalangeal 1 TUV at 60 min | 14.308134 | 11.080537
  Right proximal interphalangeal 2 TUV at 60 min | 18.710387 | 12.508548
  Right proximal interphalangeal 3 TUV at 60 min | 14.969821 | 12.831644
  Right proximal interphalangeal 4 TUV at 60 min | 18.369256 | 16.271218
  Right proximal interphalangeal 5 TUV at 60 min | 18.873772 | 16.805949
  Right wrist TUV at 60 min | 13.05914 | 10.202857
  Global TUV at 180 min: number analyzed (Participants) | 15 | 9
  Global TUV at 180 min | 355.82 | 287.80
  Left metacarpophalangeal 1 TUV at 180 min | 19.4363 | 12.081512
  Left metacarpophalangeal 2 TUV at 180 min | 21.914899 | 19.814146
  Left metacarpophalangeal 3 TUV at 180 min | 24.269644 | 15.786226
  Left metacarpophalangeal 4 TUV at 180 min | 23.438328 | 17.776583
  Left metacarpophalangeal 5 TUV at 180 min | 21.045602 | 14.647724
  Left proximal interphalangeal 1 TUV at 180 min | 18.335106 | 15.40672
  Left proximal interphalangeal 2 TUV at 180 min | 19.144279 | 10.324402
  Left proximal interphalangeal 3 TUV at 180 min | 16.707115 | 11.347808
  Left proximal interphalangeal 4 TUV at 180 min | 20.968296 | 11.384086
  Left proximal interphalangeal 5 TUV at 180 min | 15.155009 | 12.16714
  Left wrist TUV at 180 min | 17.46611 | 10.10065
  Right metacarpophalangeal 1 TUV at 180 min | 18.333323 | 12.726762
  Right metacarpophalangeal 2 TUV at 180 min | 19.876281 | 16.017255
  Right metacarpophalangeal 3 TUV at 180 min | 19.314268 | 19.791295
  Right metacarpophalangeal 4 TUV at 180 min | 21.176376 | 18.332795
  Right metacarpophalangeal 5 TUV at 180 min | 21.480266 | 13.444692
  Right proximal interphalangeal 1 TUV at 180 min | 16.290041 | 10.408102
  Right proximal interphalangeal 2 TUV at 180 min | 18.330801 | 11.916304
  Right proximal interphalangeal 3 TUV at 180 min | 17.515896 | 10.748883
  Right proximal interphalangeal 4 TUV at 180 min | 20.621393 | 16.172441
  Right proximal interphalangeal 5 TUV at 180 min | 18.927298 | 14.872591
  Right wrist TUV at 180 min | 16.823037 | 10.559086

3. Primary Outcome: Arm 3: Correlation of ΔTUVglobal[5w] and Response to Therapy
Description: The Kendall rank correlation of the change in global TUV from baseline to 5 weeks (ΔTUVglobal[5w]) and response to new anti-TNFα bDMARD therapy defined by the change from baseline of CDAI to 12 ± 1 weeks and 24 ± 1 weeks (ΔCDAI12w and ΔCDAI24w).• The Kendall rank correlation of ΔTUVglobal[5w] and response to new anti-TNFα bDMARD therapy from baseline to 12 ± 1 weeks and 24 ± 1 weeks defined by ACR Response Criteria (ΔACR12w and ΔACR24w)
Time Frame: Imaging (60 minutes after tilmanocept injection) on Day 0 and at 5 weeks after new therapy initiation; Assessment of CDAI and ACR Response Criteria at 12 and 24 weeks after new therapy initiation.
Population: All Arm 3 subjects with data at the specified timepoint (Week 12 or Week 24)
Measure: Number (95% Confidence Interval); unit: Kendall rank correlation
Groups:
- RA Subjects Who Are Candidates for Initiation of a New Anti-TNFα Therapy: Arm 3 included clinically diagnosed RA subjects on stable treatment who were candidates for new anti-TNFα therapy. Arm 3 assessed the efficacy of global TUVs, obtained before and after initiation of a new anti-TNFα therapy, to predict future clinical responsiveness to the new therapy.
  Tc99m-tilmanocept: Tilmanocept is a radiotracer that accumulates in macrophages by binding to a mannose binding receptor that resides on the surface.
Arm/Group | RA Subjects Who Are Candidates for Initiation of a New Anti-TNFα Therapy
Number analyzed (Participants) | 29
Kendall rank correlation
  ΔTUVglobal[5w] and ΔCDAI12w (overall) - Reader 1 | 0.248 [0.003 to 0.494]
  ΔTUVglobal[5w] and ΔCDAI12w (overall) - Reader 2 | 0.238 [0.002 to 0.474]
  ΔTUVglobal[5w] and ΔCDAI24w (overall) - Reader 1: number analyzed (Participants) | 27
  ΔTUVglobal[5w] and ΔCDAI24w (overall) - Reader 1 | 0.115 [-0.221 to 0.452]
  ΔTUVglobal[5w] and ΔCDAI24w (overall) - Reader 2: number analyzed (Participants) | 27
  ΔTUVglobal[5w] and ΔCDAI24w (overall) - Reader 2 | 0.121 [-0.207 to 0.449]
  ΔTUVglobal[5w] and ΔACR12w (Swollen Joint Count) - Reader 1 | 0.165 [-0.077 to 0.407]
  ΔTUVglobal[5w] and ΔACR12w (Swollen Joint Count) - Reader 2 | 0.154 [-0.096 to 0.405]
  ΔTUVglobal[5w] and ACR24w (Swollen Joint Count) - Reader 1: number analyzed (Participants) | 27
  ΔTUVglobal[5w] and ACR24w (Swollen Joint Count) - Reader 1 | 0.226 [-0.024 to 0.476]
  ΔTUVglobal[5w] and ΔACR24w (Swollen Joint Count) - Reader 2: number analyzed (Participants) | 27
  ΔTUVglobal[5w] and ΔACR24w (Swollen Joint Count) - Reader 2 | 0.235 [-0.013 to 0.483]
  ΔTUVglobal[5w] and ΔACR12w (Tender Joint Count) - Reader 1 | 0.119 [-0.152 to 0.389]
  ΔTUVglobal[5w] and ΔACR12w (Tender Joint Count) - Reader 2 | 0.138 [-0.124 to 0.399]
  ΔTUVglobal[5w] and ΔACR24w (Tender Joint Count) - Reader 1: number analyzed (Participants) | 27
  ΔTUVglobal[5w] and ΔACR24w (Tender Joint Count) - Reader 1 | 0.161 [-0.146 to 0.469]
  ΔTUVglobal[5w] and ΔACR24w (Tender Joint Count) - Reader 2: number analyzed (Participants) | 27
  ΔTUVglobal[5w] and ΔACR24w (Tender Joint Count) - Reader 2 | 0.194 [-0.110 to 0.499]
  ΔTUVglobal[5w] and ΔACR12w (ESR) - Reader 1: number analyzed (Participants) | 28
  ΔTUVglobal[5w] and ΔACR12w (ESR) - Reader 1 | -0.199 [-0.506 to 0.107]
  ΔTUVglobal[5w] and ΔACR12w (ESR) - Reader 2: number analyzed (Participants) | 28
  ΔTUVglobal[5w] and ΔACR12w (ESR) - Reader 2 | -0.110 [-0.412 to 0.192]
  ΔTUVglobal[5w] and ΔACR24w (ESR) - Reader 1: number analyzed (Participants) | 26
  ΔTUVglobal[5w] and ΔACR24w (ESR) - Reader 1 | -0.267 [-0.588 to 0.053]
  ΔTUVglobal[5w] and ΔACR24w (ESR) - Reader 2: number analyzed (Participants) | 26
  ΔTUVglobal[5w] and ΔACR24w (ESR) - Reader 2 | -0.186 [-0.493 to 0.121]
  ΔTUVglobal[5w] and ΔACR12w (VAS Pain Scale) - Reader 1 | 0.110 [-0.153 to 0.374]
  ΔTUVglobal[5w] and ΔACR12w (VAS Pain Scale) - Reader 2 | 0.105 [-0.153 to 0.362]
  ΔTUVglobal[5w] and ΔACR24w (VAS Pain Scale) - Reader 1: number analyzed (Participants) | 27
  ΔTUVglobal[5w] and ΔACR24w (VAS Pain Scale) - Reader 1 | -0.125 [-0.447 to 0.197]
  ΔTUVglobal[5w] and ΔACR24w (VAS Pain Scale) - Reader 2: number analyzed (Participants) | 27
  ΔTUVglobal[5w] and ΔACR24w (VAS Pain Scale) - Reader 2 | -0.121 [-0.433 to 0.190]
  ΔTUVglobal[5w] and ΔACR12w (Patient's Global Assessment) - Reader 1 | 0.299 [0.108 to 0.490]
  ΔTUVglobal[5w] and ΔACR12w (Patient's Global Assessment) - Reader 2 | 0.261 [0.037 to 0.484]
  ΔTUVglobal[5w] and ΔACR24w (Patient's Global Assessment) - Reader 1: number analyzed (Participants) | 27
  ΔTUVglobal[5w] and ΔACR24w (Patient's Global Assessment) - Reader 1 | 0.051 [-0.257 to 0.359]
  ΔTUVglobal[5w] and ΔACR24w (Patient's Global Assessment) - Reader 2: number analyzed (Participants) | 27
  ΔTUVglobal[5w] and ΔACR24w (Patient's Global Assessment) - Reader 2 | 0.070 [-0.226 to 0.366]
  ΔTUVglobal[5w] and ΔACR12w (Physician's Global Assessment) - Reader 1 | 0.137 [-0.090 to 0.365]
  ΔTUVglobal[5w] and ΔACR12w (Physician's Global Assessment) - Reader 2 | 0.115 [-0.117 to 0.348]
  ΔTUVglobal[5w] and ΔACR24w (Physician's Global Assessment) - Reader 1: number analyzed (Participants) | 27
  ΔTUVglobal[5w] and ΔACR24w (Physician's Global Assessment) - Reader 1 | -0.057 [-0.349 to 0.234]
  ΔTUVglobal[5w] and ΔACR24w (Physician's Global Assessment) - Reader 2: number analyzed (Participants) | 27
  ΔTUVglobal[5w] and ΔACR24w (Physician's Global Assessment) - Reader 2 | -0.032 [-0.323 to 0.259]
  ΔTUVglobal[5w] and ΔACR12w (HAQ-DI Score) - Reader 1 | 0.025 [-0.237 to 0.286]
  ΔTUVglobal[5w] and ΔACR12w (HAQ-DI Score) - Reader 2 | 0.083 [-0.167 to 0.333]
  ΔTUVglobal[5w] and ΔACR24w (HAQ-DI Score) - Reader 1: number analyzed (Participants) | 27
  ΔTUVglobal[5w] and ΔACR24w (HAQ-DI Score) - Reader 1 | -0.032 [-0.339 to 0.276]
  ΔTUVglobal[5w] and ΔACR24w (HAQ-DI Score) - Reader 2: number analyzed (Participants) | 27
  ΔTUVglobal[5w] and ΔACR24w (HAQ-DI Score) - Reader 2 | 0.051 [-0.227 to 0.329]

4. Primary Outcome: Longitudinal (8-day) Variation of TUV
Description: Longitudinal (8-day) variation of TUV analyzed for each DAS28 joint, defined as the root mean square deviation (RMSD) and 95% confidence interval for the RMSD for each joint at Day 0 vs Day 8
Time Frame: Imaging (60 minutes after tilmanocept injection) on Day 0 and Day 8
Population: All Arm 2 subjects with evaluable images at Days 0 and 8
Measure: Number (95% Confidence Interval); unit: Pixel intensity
Groups:
- Arm 2 RA Subjects on Stable Therapy: Arm 2 included clinically diagnosed RA subjects on stable treatment. Arm 2 evaluated image/re-image and test re-test (i.e., repeat dose) consistency of joint-specific and global TUVs across a variety of image acquisition intervals.
  Tc99m-tilmanocept: Tilmanocept is a radiotracer that accumulates in macrophages by binding to a mannose binding receptor that resides on the surface.
Arm/Group | Arm 2 RA Subjects on Stable Therapy
Number analyzed (Participants) | 35
Pixel intensity
  Left metacarpophalangeal 1, RMSD of TUV at Day 0 vs Day 8, Reader 1, Anterior view | 0.135 [0.109 to 0.175]
  Left metacarpophalangeal 2, RMSD of TUV at Day 0 vs Day 8, Reader 1, Anterior view | 0.151 [0.122 to 0.196]
  Left metacarpophalangeal 3, RMSD of TUV at Day 0 vs Day 8, Reader 1, Anterior view | 0.221 [0.174 to 0.280]
  Left metacarpophalangeal 4, RMSD of TUV at Day 0 vs Day 8, Reader 1, Anterior view | 0.179 [0.145 to 0.234]
  Left metacarpophalangeal 5, RMSD of TUV at Day 0 vs Day 8, Reader 1, Anterior view | 0.235 [0.186 to 0.299]
  Left proximal interphalangeal 1, RMSD of TUV at Day 0 vs Day 8, Reader 1, Anterior view | 0.263 [0.213 to 0.342]
  Left proximal interphalangeal 2, RMSD of TUV at Day 0 vs Day 8, Reader 1, Anterior view | 0.198 [0.160 to 0.257]
  Left proximal interphalangeal 3, RMSD of TUV at Day 0 vs Day 8, Reader 1, Anterior view | 0.172 [0.139 to 0.224]
  Left proximal interphalangeal 4, RMSD of TUV at Day 0 vs Day 8, Reader 1, Anterior view | 0.229 [0.185 to 0.298]
  Left proximal interphalangeal 5, RMSD of TUV at Day 0 vs Day 8, Reader 1, Anterior view | 0.233 [0.181 to 0.291]
  Left wrist, RMSD of TUV at Day 0 vs Day 8, Reader 1, Anterior view | 0.107 [0.084 to 0.135]
  Right metacarpophalangeal 1, RMSD of TUV at Day 0 vs Day 8, Reader 1, Anterior view | 0.142 [0.115 to 0.185]
  Right metacarpophalangeal 2, RMSD of TUV at Day 0 vs Day 8, Reader 1, Anterior view | 0.134 [0.109 to 0.175]
  Right metacarpophalangeal 3, RMSD of TUV at Day 0 vs Day 8, Reader 1, Anterior view | 0.131 [0.106 to 0.171]
  Right metacarpophalangeal 4, RMSD of TUV at Day 0 vs Day 8, Reader 1, Anterior view | 0.208 [0.167 to 0.268]
  Right metacarpophalangeal 5, RMSD of TUV at Day 0 vs Day 8, Reader 1, Anterior view | 0.213 [0.167 to 0.269]
  Right proximal interphalangeal 1, RMSD of TUV at Day 0 vs Day 8, Reader 1, Anterior view | 0.221 [0.176 to 0.283]
  Right proximal interphalangeal 2, RMSD of TUV at Day 0 vs Day 8, Reader 1, Anterior view | 0.227 [0.182 to 0.292]
  Right proximal interphalangeal 3, RMSD of TUV at Day 0 vs Day 8, Reader 1, Anterior view | 0.212 [0.169 to 0.271]
  Right proximal interphalangeal 4, RMSD of TUV at Day 0 vs Day 8, Reader 1, Anterior view | 0.261 [0.206 to 0.332]
  Right proximal interphalangeal 5, RMSD of TUV at Day 0 vs Day 8, Reader 1, Anterior view | 0.244 [0.196 to 0.315]
  Right wrist, RMSD of TUV at Day 0 vs Day 8, Reader 1, Anterior view | 0.078 [0.063 to 0.102]
  Left metacarpophalangeal 1, RMSD of TUV at Day 0 vs Day 8, Reader 2, Anterior view | 0.180 [0.137 to 0.219]
  Left metacarpophalangeal 2, RMSD of TUV at Day 0 vs Day 8, Reader 2, Anterior view | 0.170 [0.137 to 0.221]
  Left metacarpophalangeal 3, RMSD of TUV at Day 0 vs Day 8, Reader 2, Anterior view | 0.148 [0.119 to 0.191]
  Left metacarpophalangeal 4, RMSD of TUV at Day 0 vs Day 8, Reader 2, Anterior view | 0.130 [0.104 to 0.168]
  Left metacarpophalangeal 5, RMSD of TUV at Day 0 vs Day 8, Reader 2, Anterior view | 0.180 [0.142 to 0.228]
  Left proximal interphalangeal 1, RMSD of TUV at Day 0 vs Day 8, Reader 2, Anterior view | 0.346 [0.277 to 0.445]
  Left proximal interphalangeal 2, RMSD of TUV at Day 0 vs Day 8, Reader 2, Anterior view | 0.245 [0.198 to 0.318]
  Left proximal interphalangeal 3, RMSD of TUV at Day 0 vs Day 8, Reader 2, Anterior view | 0.160 [0.129 to 0.208]
  Left proximal interphalangeal 4, RMSD of TUV at Day 0 vs Day 8, Reader 2, Anterior view | 0.202 [0.163 to 0.262]
  Left proximal interphalangeal 5, RMSD of TUV at Day 0 vs Day 8, Reader 2, Anterior view | 0.242 [0.193 to 0.310]
  Left wrist, RMSD of TUV at Day 0 vs Day 8, Reader 2, Anterior view | 0.106 [0.079 to 0.126]
  Right metacarpophalangeal 1, RMSD of TUV at Day 0 vs Day 8, Reader 2, Anterior view | 0.137 [0.109 to 0.175]
  Right metacarpophalangeal 2, RMSD of TUV at Day 0 vs Day 8, Reader 2, Anterior view | 0.120 [0.096 to 0.154]
  Right metacarpophalangeal 3, RMSD of TUV at Day 0 vs Day 8, Reader 2, Anterior view | 0.124 [0.099 to 0.160]
  Right metacarpophalangeal 4, RMSD of TUV at Day 0 vs Day 8, Reader 2, Anterior view | 0.159 [0.128 to 0.206]
  Right metacarpophalangeal 5, RMSD of TUV at Day 0 vs Day 8, Reader 2, Anterior view | 0.165 [0.133 to 0.213]
  Right proximal interphalangeal 2, RMSD of TUV at Day 0 vs Day 8, Reader 2, Anterior view | 0.237 [0.192 to 0.309]
  Right proximal interphalangeal 3, RMSD of TUV at Day 0 vs Day 8, Reader 2, Anterior view | 0.172 [0.138 to 0.222]
  Right proximal interphalangeal 4, RMSD of TUV at Day 0 vs Day 8, Reader 2, Anterior view | 0.219 [0.178 to 0.286]
  Right proximal interphalangeal 5, RMSD of TUV at Day 0 vs Day 8, Reader 2, Anterior view | 0.271 [0.215 to 0.345]
  Right wrist, RMSD of TUV at Day 0 vs Day 8, Reader 2, Anterior view | 0.084 [0.062 to 0.098]
  Left metacarpophalangeal 1, RMSD of TUV at Day 0 vs Day 8, Reader 1, Posterior view | 0.251 [0.203 to 0.326]
  Left metacarpophalangeal 2, RMSD of TUV at Day 0 vs Day 8, Reader 1, Posterior view | 0.229 [0.182 to 0.293]
  Left metacarpophalangeal 3, RMSD of TUV at Day 0 vs Day 8, Reader 1, Posterior view | 0.225 [0.180 to 0.290]
  Left metacarpophalangeal 4, RMSD of TUV at Day 0 vs Day 8, Reader 1, Posterior view | 0.224 [0.182 to 0.292]
  Left metacarpophalangeal 5, RMSD of TUV at Day 0 vs Day 8, Reader 1, Posterior view | 0.357 [0.289 to 0.465]
  Left proximal interphalangeal 1, RMSD of TUV at Day 0 vs Day 8, Reader 1, Posterior view | 0.303 [0.245 to 0.395]
  Left proximal interphalangeal 2, RMSD of TUV at Day 0 vs Day 8, Reader 1, Posterior view | 0.254 [0.199 to 0.321]
  Left proximal interphalangeal 3, RMSD of TUV at Day 0 vs Day 8, Reader 1, Posterior view | 0.251 [0.203 to 0.326]
  Left proximal interphalangeal 4, RMSD of TUV at Day 0 vs Day 8, Reader 1, Posterior view | 0.240 [0.187 to 0.300]
  Left proximal interphalangeal 5, RMSD of TUV at Day 0 vs Day 8, Reader 1, Posterior view | 0.313 [0.254 to 0.408]
  Left wrist, RMSD of TUV at Day 0 vs Day 8, Reader 1, Posterior view | 0.180 [0.146 to 0.234]
  Right metacarpophalangeal 1, RMSD of TUV at Day 0 vs Day 8, Reader 1, Posterior view | 0.288 [0.233 to 0.375]
  Right metacarpophalangeal 2, RMSD of TUV at Day 0 vs Day 8, Reader 1, Posterior view | 0.214 [0.173 to 0.278]
  Right metacarpophalangeal 3, RMSD of TUV at Day 0 vs Day 8, Reader 1, Posterior view | 0.143 [0.114 to 0.183]
  Right metacarpophalangeal 4, RMSD of TUV at Day 0 vs Day 8, Reader 1, Posterior view | 0.188 [0.149 to 0.239]
  Right metacarpophalangeal 5, RMSD of TUV at Day 0 vs Day 8, Reader 1, Posterior view | 0.247 [0.195 to 0.314]
  Right proximal interphalangeal 1, RMSD of TUV at Day 0 vs Day 8, Reader 1, Posterior view | 0.307 [0.249 to 0.400]
  Right proximal interphalangeal 2, RMSD of TUV at Day 0 vs Day 8, Reader 1, Posterior view | 0.253 [0.204 to 0.328]
  Right proximal interphalangeal 3, RMSD of TUV at Day 0 vs Day 8, Reader 1, Posterior view | 0.221 [0.178 to 0.286]
  Right proximal interphalangeal 4, RMSD of TUV at Day 0 vs Day 8, Reader 1, Posterior view | 0.246 [0.200 to 0.321]
  Right proximal interphalangeal 5, RMSD of TUV at Day 0 vs Day 8, Reader 1, Posterior view | 0.367 [0.297 to 0.477]
  Right wrist, RMSD of TUV at Day 0 vs Day 8, Reader 1, Posterior view | 0.133 [0.108 to 0.173]
  Left metacarpophalangeal 1, RMSD of TUV at Day 0 vs Day 8, Reader 2, Posterior view | 0.112 [0.087 to 0.139]
  Left metacarpophalangeal 2, RMSD of TUV at Day 0 vs Day 8, Reader 2, Posterior view | 0.112 [0.090 to 0.144]
  Left metacarpophalangeal 3, RMSD of TUV at Day 0 vs Day 8, Reader 2, Posterior view | 0.105 [0.085 to 0.136]
  Left metacarpophalangeal 4, RMSD of TUV at Day 0 vs Day 8, Reader 2, Posterior view | 0.109 [0.088 to 0.142]
  Left metacarpophalangeal 5, RMSD of TUV at Day 0 vs Day 8, Reader 2, Posterior view | 0.152 [0.123 to 0.198]
  Left proximal interphalangeal 1, RMSD of TUV at Day 0 vs Day 8, Reader 2, Posterior view | 0.227 [0.180 to 0.290]
  Left proximal interphalangeal 2, RMSD of TUV at Day 0 vs Day 8, Reader 2, Posterior view | 0.133 [0.108 to 0.173]
  Left proximal interphalangeal 3, RMSD of TUV at Day 0 vs Day 8, Reader 2, Posterior view | 0.183 [0.147 to 0.237]
  Left proximal interphalangeal 4, RMSD of TUV at Day 0 vs Day 8, Reader 2, Posterior view | 0.205 [0.161 to 0.259]
  Left proximal interphalangeal 5, RMSD of TUV at Day 0 vs Day 8, Reader 2, Posterior view | 0.281 [0.221 to 0.356]
  Left wrist, RMSD of TUV at Day 0 vs Day 8, Reader 2, Posterior view | 0.081 [0.062 to 0.099]
  Right metacarpophalangeal 1, RMSD of TUV at Day 0 vs Day 8, Reader 2, Posterior view | 0.149 [0.120 to 0.194]
  Right metacarpophalangeal 2, RMSD of TUV at Day 0 vs Day 8, Reader 2, Posterior view | 0.141 [0.111 to 0.179]
  Right metacarpophalangeal 3, RMSD of TUV at Day 0 vs Day 8, Reader 2, Posterior view | 0.132 [0.107 to 0.173]
  Right metacarpophalangeal 4, RMSD of TUV at Day 0 vs Day 8, Reader 2, Posterior view | 0.137 [0.109 to 0.175]
  Right metacarpophalangeal 5, RMSD of TUV at Day 0 vs Day 8, Reader 2, Posterior view | 0.165 [0.134 to 0.215]
  Right proximal interphalangeal 1, RMSD of TUV at Day 0 vs Day 8, Reader 2, Posterior view | 1.834 [1.471 to 2.365]
  Right proximal interphalangeal 2, RMSD of TUV at Day 0 vs Day 8, Reader 2, Posterior view | 0.178 [0.144 to 0.231]
  Right proximal interphalangeal 3, RMSD of TUV at Day 0 vs Day 8, Reader 2, Posterior view | 0.199 [0.160 to 0.257]
  Right proximal interphalangeal 4, RMSD of TUV at Day 0 vs Day 8, Reader 2, Posterior view | 0.200 [0.162 to 0.260]
  Right proximal interphalangeal 5, RMSD of TUV at Day 0 vs Day 8, Reader 2, Posterior view | 0.215 [0.174 to 0.279]
  Right wrist, RMSD of TUV at Day 0 vs Day 8, Reader 2, Posterior view | 0.081 [0.065 to 0.104]

5. Secondary Outcome: Arm 1 Normal Ranges of TUVjoint
Description: The normal range of tilmanocept uptake values (TUVs) in hand and wrist joints of healthy control subjects, expressed as the mean and standard deviation. TUV is defined as the average pixel intensity of the region of interest (hand or wrist joint) divided by the average pixel intensity of the reference region (includes the region from one wrist region of interest diameter above the wrist region of interest down to the fingertips)
Time Frame: Images obtained 60 minutes after tilmanocept injection on Day 0.
Population: Healthy control subjects with evaluable scans. Unevaluable scans included those with poor hand placement/positioning and low signal (overlapping with background) in most of the fingers.
Measure: Mean (Standard Deviation); unit: Pixel intensity
Groups:
- Subjects Free of Inflammatory Disease: Arm 1 included inflammatory-disease-free HCs. Arm 1 evaluated image/re-image consistency (repeatability and stability) of joint-specific and global TUVs across a variety of image acquisition intervals and collected normative HC data.
  Tc99m-tilmanocept: Tilmanocept is a radiotracer that accumulates in macrophages by binding to a mannose binding receptor that resides on the surface.
Arm/Group | Subjects Free of Inflammatory Disease
Number analyzed (Participants) | 29
Pixel intensity
  Left Metacarpophalangeal 1, Anterior View, Reader 1 | 1.01 (0.213)
  Left Metacarpophalangeal 1, Anterior View, Reader 2 | 1.20 (0.257)
  Left Metacarpophalangeal 1, Posterior View, Reader 1 | 1.05 (0.185)
  Left Metacarpophalangeal 1, Posterior View, Reader 2 | 1.33 (0.200)
  Left Metacarpophalangeal 2, Anterior View, Reader 1 | 0.85 (0.169)
  Left Metacarpophalangeal 2, Anterior View, Reader 2 | 0.92 (0.180)
  Left Metacarpophalangeal 2, Posterior View, Reader 1 | 0.86 (0.158)
  Left Metacarpophalangeal 2, Posterior View, Reader 2 | 1.00 (0.170)
  Left Metacarpophalangeal 3, Anterior View, Reader 1 | 0.79 (0.158)
  Left Metacarpophalangeal 3, Anterior View, Reader 2 | 0.90 (0.197)
  Left Metacarpophalangeal 3, Posterior View, Reader 1 | 0.86 (0.186)
  Left Metacarpophalangeal 3, Posterior View, Reader 2 | 1.04 (0.174)
  Left Metacarpophalangeal 4, Anterior View, Reader 1 | 0.77 (0.192)
  Left Metacarpophalangeal 4, Anterior View, Reader 2 | 0.90 (0.201)
  Left Metacarpophalangeal 4, Posterior View, Reader 1 | 0.80 (0.144)
  Left Metacarpophalangeal 4, Posterior View, Reader 2 | 1.01 (0.161)
  Left Metacarpophalangeal 5, Anterior View, Reader 1 | 0.73 (0.186)
  Left Metacarpophalangeal 5, Anterior View, Reader 2 | 0.82 (0.189)
  Left Metacarpophalangeal 5, Posterior View, Reader 1 | 0.80 (0.162)
  Left Metacarpophalangeal 5, Posterior View, Reader 2 | 0.92 (0.169)
  Left Proximal Interphalangeal 1, Anterior View, Reader 1 | 0.75 (0.158)
  Left Proximal Interphalangeal 1, Anterior View, Reader 2 | 0.89 (0.192)
  Left Proximal Interphalangeal 1, Posterior View, Reader 1 | 0.79 (0.175)
  Left Proximal Interphalangeal 1, Posterior View, Reader 2 | 0.93 (0.166)
  Left Proximal Interphalangeal 2, Anterior View, Reader 1 | 0.71 (0.170)
  Left Proximal Interphalangeal 2, Anterior View, Reader 2 | 0.77 (0.179)
  Left Proximal Interphalangeal 2, Posterior View, Reader 1 | 0.68 (0.129)
  Left Proximal Interphalangeal 2, Posterior View, Reader 2 | 0.79 (0.155)
  Left Proximal Interphalangeal 3, Anterior View, Reader 1 | 0.70 (0.184)
  Left Proximal Interphalangeal 3, Anterior View, Reader 2 | 0.73 (0.192)
  Left Proximal Interphalangeal 3, Posterior View, Reader 1 | 0.69 (0.126)
  Left Proximal Interphalangeal 3, Posterior View, Reader 2 | 0.82 (0.146)
  Left Proximal Interphalangeal 4, Anterior View, Reader 1 | 0.66 (0.143)
  Left Proximal Interphalangeal 4, Anterior View, Reader 2 | 0.72 (0.167)
  Left Proximal Interphalangeal 4, Posterior View, Reader 1 | 0.64 (0.128)
  Left Proximal Interphalangeal 4, Posterior View, Reader 2 | 0.75 (0.156)
  Left Proximal Interphalangeal 5, Anterior View, Reader 1 | 0.59 (0.147)
  Left Proximal Interphalangeal 5, Anterior View, Reader 2 | 0.66 (0.141)
  Left Proximal Interphalangeal 5, Posterior View, Reader 1 | 0.59 (0.124)
  Left Proximal Interphalangeal 5, Posterior View, Reader 2 | 0.69 (0.135)
  Left Wrist, Anterior View, Reader 1 | 1.32 (0.229)
  Left Wrist, Anterior View, Reader 2 | 1.48 (0.243)
  Left Wrist, Posterior View, Reader 1 | 1.40 (0.183)
  Left Wrist, Posterior View, Reader 2 | 1.66 (0.180)
  Right Metacarpophalangeal 1, Anterior View, Reader 1 | 0.98 (0.185)
  Right Metacarpophalangeal 1, Anterior View, Reader 2 | 1.17 (0.244)
  Right Metacarpophalangeal 1, Posterior View, Reader 1 | 1.04 (0.190)
  Right Metacarpophalangeal 1, Posterior View, Reader 2 | 1.29 (0.297)
  Right Metacarpophalangeal 2, Anterior View, Reader 1 | 0.87 (0.180)
  Right Metacarpophalangeal 2, Anterior View, Reader 2 | 0.88 (0.181)
  Right Metacarpophalangeal 2, Posterior View, Reader 1 | 0.94 (0.206)
  Right Metacarpophalangeal 2, Posterior View, Reader 2 | 1.00 (0.182)
  Right Metacarpophalangeal 3, Anterior View, Reader 1 | 0.83 (0.176)
  Right Metacarpophalangeal 3, Anterior View, Reader 2 | 0.91 (0.191)
  Right Metacarpophalangeal 3, Posterior View, Reader 1 | 0.86 (0.143)
  Right Metacarpophalangeal 3, Posterior View, Reader 2 | 1.02 (0.189)
  Right Metacarpophalangeal 4, Anterior View, Reader 1 | 0.83 (0.214)
  Right Metacarpophalangeal 4, Anterior View, Reader 2 | 0.94 (0.216)
  Right Metacarpophalangeal 4, Posterior View, Reader 1 | 0.83 (0.141)
  Right Metacarpophalangeal 4, Posterior View, Reader 2 | 1.02 (0.199)
  Right Metacarpophalangeal 5, Anterior View, Reader 1 | 0.74 (0.174)
  Right Metacarpophalangeal 5, Anterior View, Reader 2 | 0.86 (0.212)
  Right Metacarpophalangeal 5, Posterior View, Reader 1 | 0.78 (0.156)
  Right Metacarpophalangeal 5, Posterior View, Reader 2 | 0.96 (0.200)
  Right Proximal Interphalangeal 1, Anterior View, Reader 1 | 0.79 (0.162)
  Right Proximal Interphalangeal 1, Anterior View, Reader 2 | 0.89 (0.198)
  Right Proximal Interphalangeal 1, Posterior View, Reader 1 | 0.80 (0.161)
  Right Proximal Interphalangeal 1, Posterior View, Reader 2 | 0.95 (0.155)
  Right Proximal Interphalangeal 2, Anterior View, Reader 1 | 0.68 (0.140)
  Right Proximal Interphalangeal 2, Anterior View, Reader 2 | 0.75 (0.159)
  Right Proximal Interphalangeal 2, Posterior View, Reader 1 | 0.73 (0.114)
  Right Proximal Interphalangeal 2, Posterior View, Reader 2 | 0.79 (0.129)
  Right Proximal Interphalangeal 3, Anterior View, Reader 1 | 0.66 (0.164)
  Right Proximal Interphalangeal 3, Anterior View, Reader 2 | 0.73 (0.183)
  Right Proximal Interphalangeal 3, Posterior View, Reader 1 | 0.71 (0.118)
  Right Proximal Interphalangeal 3, Posterior View, Reader 2 | 0.80 (0.139)
  Right Proximal Interphalangeal 4, Anterior View, Reader 1 | 0.67 (0.196)
  Right Proximal Interphalangeal 4, Anterior View, Reader 2 | 0.73 (0.172)
  Right Proximal Interphalangeal 4, Posterior View, Reader 1 | 0.65 (0.132)
  Right Proximal Interphalangeal 4, Posterior View, Reader 2 | 0.73 (0.142)
  Right Proximal Interphalangeal 5, Anterior View, Reader 1 | 0.58 (0.141)
  Right Proximal Interphalangeal 5, Anterior View, Reader 2 | 0.66 (0.135)
  Right Proximal Interphalangeal 5, Posterior View, Reader 1 | 0.55 (0.093)
  Right Proximal Interphalangeal 5, Posterior View, Reader 2 | 0.66 (0.122)
  Right Wrist, Anterior View, Reader 1 | 1.35 (0.221)
  Right Wrist, Anterior View, Reader 2 | 1.51 (0.253)
  Right Wrist, Posterior View, Reader 1 | 1.41 (0.188)
  Right Wrist, Posterior View, Reader 2 | 1.65 (0.264)

6. Secondary Outcome: Qualitative Evaluations of SPECT/CT as an Indication of Bone Involvement Rather Than Localization Within the Synovial Space in the Hands and Wrists of Arm 2 Subjects
Description: Percent of Arm 2 subjects who had SPECT/CT scans who were determined to have bone involvement rather than localization within the synovial space of the hands and wrists
Time Frame: A SPECT/CT scan was performed at approximately 210 minutes after the tilmanocept injection on Day 8 of the trial.
Population: All Arm 2 subjects who received SPECT/CT scan
Measure: Number; unit: Percent of participants
Arm/Group | Arm 2 RA Subjects on Stable Therapy
Number analyzed (Participants) | 20
Percent of participants | 0

7. Secondary Outcome: Arm 3 (Correlation of TUVglobal[Baseline] and Response to Therapy)
Description: The correlation of the TUVglobal[baseline] and response to new anti-TNFα bDMARD therapy defined by the change from baseline (CFB) of CDAI to 12 ± 1 weeks and 24 ± 1 weeks (ΔCDAI12w and ΔCDAI24w, respectively) and by ACR Response Criteria (ACR12w and ACR24w, respectively).
Time Frame: Images were obtained 60 minutes after tilmanocept injection on Day 0. New anti-TNFα therapy was initiated after completion of Day 0 procedures. CDAI and ACR were assessed on Day 0 and again 12 and 24 weeks after initiation of new anti-TNFα therapy.
Population: All Arm 3 subjects with data at the specified timepoint (Week 12 or Week 24)
Measure: Number (95% Confidence Interval); unit: Kendall rank correlation
Arm/Group | RA Subjects Who Are Candidates for Initiation of a New Anti-TNFα Therapy
Number analyzed (Participants) | 29
Kendall rank correlation
  TUVglobal[baseline] and ΔCDAI12w (overall) - Reader 1: number analyzed (Participants) | 28
  TUVglobal[baseline] and ΔCDAI12w (overall) - Reader 1 | -0.045 [-0.320 to 0.229]
  TUVglobal[baseline] and ΔCDAI24w (overall) - Reader 1: number analyzed (Participants) | 27
  TUVglobal[baseline] and ΔCDAI24w (overall) - Reader 1 | 0.072 [-0.215 to 0.359]
  TUVglobal[baseline] and ΔACR12w (Swollen Joint Count) - Reader 1 | -0.100 [-0.387 to 0.186]
  TUVglobal[baseline] and ΔACR24w (Swollen Joint Count) - Reader 1: number analyzed (Participants) | 27
  TUVglobal[baseline] and ΔACR24w (Swollen Joint Count) - Reader 1 | -0.067 [-0.391 to 0.258]
  TUVglobal[baseline] and ΔACR12w (Tender Joint Count) - Reader 1 | -0.086 [-0.317 to 0.144]
  TUVglobal[baseline] and ΔACR24w (Tender Joint Count) - Reader 1: number analyzed (Participants) | 27
  TUVglobal[baseline] and ΔACR24w (Tender Joint Count) - Reader 1 | 0.130 [-0.171 to 0.430]
  TUVglobal[baseline] and ΔACR12w (ESR) - Reader 1: number analyzed (Participants) | 28
  TUVglobal[baseline] and ΔACR12w (ESR) - Reader 1 | -0.176 [-0.473 to 0.120]
  TUVglobal[baseline] and ΔACR24w (ESR) - Reader 1: number analyzed (Participants) | 26
  TUVglobal[baseline] and ΔACR24w (ESR) - Reader 1 | -0.261 [-0.471 to -0.051]
  TUVglobal[baseline] and ΔACR12w (VAS Pain Scale) - Reader 1 | -0.099 [-0.292 to 0.093]
  TUVglobal[baseline] and ΔACR24w (VAS Pain Scale) - Reader 1: number analyzed (Participants) | 27
  TUVglobal[baseline] and ΔACR24w (VAS Pain Scale) - Reader 1 | -0.062 [-0.303 to 0.178]
  TUVglobal[baseline] and ΔACR12w (Patient's Global Assessment) - Reader 1 | -0.096 [-0.393 to 0.201]
  TUVglobal[baseline] and ΔACR24w (Patient's Global Assessment) - Reader 1: number analyzed (Participants) | 27
  TUVglobal[baseline] and ΔACR24w (Patient's Global Assessment) - Reader 1 | -0.070 [-0.323 to 0.183]
  TUVglobal[baseline] and ΔACR12w (Physician's Global Assessment) - Reader 1 | 0.121 [-0.212 to 0.454]
  TUVglobal[baseline] and ΔACR24w (Physician's Global Assessment) - Reader 1: number analyzed (Participants) | 27
  TUVglobal[baseline] and ΔACR24w (Physician's Global Assessment) - Reader 1 | 0.057 [-0.254 to 0.369]
  TUVglobal[baseline] and ΔCDAI12w (overall) - Reader 2 | -0.029 [-0.299 to 0.241]
  TUVglobal[baseline] and ΔCDAI24w (overall) - Reader 2: number analyzed (Participants) | 27
  TUVglobal[baseline] and ΔCDAI24w (overall) - Reader 2 | 0.109 [-0.176 to 0.393]
  TUVglobal[baseline] and ΔACR12w (Swollen Joint Count) - Reader 2 | -0.073 [-0.356 to 0.210]
  TUVglobal[baseline] and ΔACR24w (Swollen Joint Count) - Reader 2: number analyzed (Participants) | 27
  TUVglobal[baseline] and ΔACR24w (Swollen Joint Count) - Reader 2 | -0.025 [-0.349 to 0.298]
  TUVglobal[baseline] and ΔACR12w (Tender Joint Count) - Reader 2 | -0.057 [-0.298 to 0.184]
  TUVglobal[baseline] and ΔACR24w (Tender Joint Count) - Reader 2: number analyzed (Participants) | 27
  TUVglobal[baseline] and ΔACR24w (Tender Joint Count) - Reader 2 | 0.175 [-0.131 to 0.482]
  TUVglobal[baseline] and ΔACR12w (ESR) - Reader 2: number analyzed (Participants) | 28
  TUVglobal[baseline] and ΔACR12w (ESR) - Reader 2 | -0.145 [-0.454 to 0.165]
  TUVglobal[baseline] and ΔACR24w (ESR) - Reader 2: number analyzed (Participants) | 26
  TUVglobal[baseline] and ΔACR24w (ESR) - Reader 2 | -0.234 [-0.468 to 0.001]
  TUVglobal[baseline] and ΔACR12w (VAS Pain Scale) - Reader 2 | -0.110 [-0.303 to 0.083]
  TUVglobal[baseline] and ΔACR24w (VAS Pain Scale) - Reader 2: number analyzed (Participants) | 27
  TUVglobal[baseline] and ΔACR24w (VAS Pain Scale) - Reader 2 | -0.028 [-0.263 to 0.207]
  TUVglobal[baseline] and ΔACR12w (Patient's Global Assessment) - Reader 2 | -0.096 [-0.384 to 0.192]
  TUVglobal[baseline] and ΔACR24w (Patient's Global Assessment) - Reader 2: number analyzed (Participants) | 27
  TUVglobal[baseline] and ΔACR24w (Patient's Global Assessment) - Reader 2 | -0.038 [-0.295 to 0.219]
  TUVglobal[baseline] and ΔACR12w (Physician's Global Assessment) - Reader 2 | 0.110 [-0.223 to 0.443]
  TUVglobal[baseline] and ΔACR24w (Physician's Global Assessment) - Reader 2: number analyzed (Participants) | 27
  TUVglobal[baseline] and ΔACR24w (Physician's Global Assessment) - Reader 2 | 0.064 [-0.251 to 0.379]

ADVERSE EVENTS:
Time Frame: Untoward medical events beginning on Visit 2 (Day 0) until the final visit (variable per arm) were reported as adverse events. For subjects in Arms 1 and 2, the final visit (Visit 5) occurred on Day 8 to 12. For subjects in Arm 3, the final visit (Visit 9) occurred on Week 24 to 26.
Groups:
- Subjects Free of Inflammatory Disease: Arm 1 included inflammatory-disease-free HCs. Arm 1 evaluated image/re-image consistency (repeatability and stability) of joint-specific and global TUVs across a variety of image acquisition intervals and collect normative HC data.
  Tc99m-tilmanocept: Tilmanocept is a radiotracer that accumulates in macrophages by binding to a mannose binding receptor that resides on the surface.
- RA Subjects on Stable Therapy: Arm 2 included clinically diagnosed RA subjects on stable treatment. Arm 2 evaluated image/re-image and test re-test (i.e., repeat dose) consistency of joint-specific and global TUVs across a variety of image acquisition intervals.
  Tc99m-tilmanocept: Tilmanocept is a radiotracer that accumulates in macrophages by binding to a mannose binding receptor that resides on the surface.
Arm/Group | Subjects Free of Inflammatory Disease | RA Subjects on Stable Therapy | RA Subjects Who Are Candidates for Initiation of a New Anti-TNFα Therapy
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/41 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/41 | 2/31
Other Adverse Events (participants affected / at risk) | 0/44 | 8/41 | 9/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects Free of Inflammatory Disease (N=44) | RA Subjects on Stable Therapy (N=41) | RA Subjects Who Are Candidates for Initiation of a New Anti-TNFα Therapy (N=31)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects Free of Inflammatory Disease (N=44) | RA Subjects on Stable Therapy (N=41) | RA Subjects Who Are Candidates for Initiation of a New Anti-TNFα Therapy (N=31)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1)
Vitreous floaters (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Hordeolum (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Chest pain (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site bruising (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Corona virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Acute coronary syndrome (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-02-02): https://cdn.clinicaltrials.gov/large-docs/36/NCT03938636/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-06): https://cdn.clinicaltrials.gov/large-docs/36/NCT03938636/SAP_001.pdf